CLINICAL TRIAL: NCT01220349
Title: Early Detection of Diabetic Cardiomyopathy by Analysis of Myocardial Deformations by Two-dimensional Speckle Tracking Strain Echocardiography and Relationship to Micro-angiopathy
Brief Title: Alteration of Myocardial Deformations in Diabetes: Relationship to Micro-angiopathy
Acronym: ECHO-DIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2009/27
Record Dates: First submitted 2010-10-07; First posted 2010-10-13 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echocardiographic 2D strain analysis (Experimental)
  Interventions: Device: Echocardiographic 2D strain analysis

INTERVENTIONS:
Device: Echocardiographic 2D strain analysis — Conventional transthoracic echocardiography with acquisitions for strain analysis by speckle tracking (2D strain)

SUMMARY:
Despite careful monitoring of patients with diabetes, it is so far difficult to predict the occurrence of cardiac events in the evolution. As shown by various studies conducted in patients with diabetes, cardiac involvement can be detected by abnormalities of diastolic or systolic functions using non-invasive investigations such as echocardiography. For 4 years, the evaluation technique of myocardial deformations by two-dimensional speckle tracking strain by echocardiography is the subject of high hopes in the earlier detection of still asymptomatic cardiomyopathies. In the present study, the investigators hypothesized that this technique would improve the detection of myocardial contraction abnormalities in patients with insulin-dependent diabetes mellitus (IDDM), and would establish their association with micro-angiopathy, frequently encountered in these patients.

DETAILED DESCRIPTION:
This is a single center case-control study based on routine care, designed to recruit patients with type 1 diabetes mellitus free from any other myocardiopathy. The inclusion will take place over a period of 24 months. No monitoring of patients (no follow-up) is provided under this protocol. The analysis will focus on the combination of the left ventricle myocardial deformations alteration revealed by the echocardiographic 2D strain analysis (< 18% in absolute value), with the existence of micro-angiopathy in type 1 diabetes mellitus patients with preserved left ventricular ejection fraction ( ≥ 60%).

Two hundred subjects with type 1 diabetes mellitus will be recruited: 100 subjects with impaired left ventricular myocardial deformation by 2D strain analysis (< 18% in absolute value), constituting the 'cases' group and 100 subjects without alteration in myocardial deformation (global strain ≥ 18%).

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 45 years
* with diagnosed Type 1 diabetes mellitus (with or without complications or peripheric vascular micro-angiopathy)
* having a negative myocardial ischemic test (exercise echocardiography) in the previous month inclusion

Exclusion Criteria:

* Known or suspected coronary artery disease
* atrial fibrillation
* hypertension
* moderate to severe valvular disease
* sequelae of myocardial infarction
* secondary or primary cardiomyopathy
* myocardial conduction abnormalities
* pregnancy or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Measurement of the alteration of left ventricular myocardial strain (≤ 18% in absolute value) by echocardiography and the relationship to micro-angiopathy. | Inclusion : Day 1

SECONDARY OUTCOMES:
Analyses of this association (alteration of myocardial strain and micro-angiopathy) in relation with the duration of diabetes, and other co-factors such as dyslipidemia, unstable diabetes, and coexisting macro-angiopathy. | Inclusion : Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Patricia REANT, MD-PhD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Hôpital Cardiologique du Haut-Lévêque, Service de Cardiologie et Maladies Vasculaires, Pessac, France